CLINICAL TRIAL: NCT03331627
Title: A Phase III Multicenter, Double-blind, Placebo-controlled, Study Evaluating the Safety, and Efficacy of STR001 Treatment in Adults With Sudden Sensorineural Hearing Loss
Brief Title: Safety and Efficacy of STR001-IT and STR001-ER in Patients With SSHL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Strekin AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-000242-22
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2019-04

CONDITIONS: Acute Hearing Loss

STUDY DESIGN:
Intervention Model Description: 1. intratympanic gel injection followed by 12 weeks oral treatment
  2. intratympanic gel injection followed by 12 weeks oral treatment placebo
  3. intratympanic gel injection placebo followed by 12 weeks oral treatment placebo
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- STR001-IT/STR001-ER (Active Comparator)
  Interventions: Drug: STR001-IT and STR001-ER
- STR001-IT/STR001-ER Placebo (Active Comparator)
  Interventions: Drug: STR001-IT and STR001-ER
- STR001-IT placebo/STR001- ER placebo (Placebo Comparator)
  Interventions: Drug: STR001-IT and STR001-ER

INTERVENTIONS:
Drug: STR001-IT and STR001-ER — STR001-IT intrataympanic injection and STR001-ER tablet

SUMMARY:
a multicenter, double-blind, placebo-controlled study in patients with Sudden Sensorineural Hearing Loss (SSHL). Patients will be treated with STR001 thermogel (STR001-IT) / STR001 tablets (STR001-ER) and corresponding Placebo on top of standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 18
2. Patients with a SSHL within 96 hours of its perception
3. Sudden Sensorineural Hearing Loss including

   1. idiopathic unilateral Sudden Sensorineural Hearing Loss or
   2. acute uni- or bilateral acoustic trauma-induced Sudden Sensorineural Hearing Loss

Exclusion Criteria:

1. Patients with a history of Meniere's Disease
2. Patients with a hearing threshold above 100 dB across at least 6 frequencies
3. Patients with endolymphatic, hydrops or history of fluctuating hearing loss
4. Patients with suspected perilymph fistula, membrane rupture, retrocochlear lesions or a barotrauma
5. Patients with an air-bone gap of ≥ 20 dB in 3 contiguous frequencies at baseline
6. Previous SSHL incident at the same ear
7. Patients with acute or chronic otitis media or otitis externa.
8. Patients with congenital hearing loss
9. Patients with known hypersensitivity to pioglitazone, other thiazolidindiones or any formulation component
10. Use of thiazolidinedione (e.g. pioglitazone, rosiglitazone) in the last 6 months prior to baseline
11. Any use of CYP450 2C8 inducers (e.g. rifampicine)
12. Fibrates (e.g. gemfibrozil, fenofibrate) in the last 6 months prior to baseline
13. Patients where oral administration of pioglitazone is contraindicated (i.e. cardiac failure or history of cardiac failure (NYHA stages I to IV), hepatic impairment, diabetic ketoacidosis, current bladder cancer or a history of bladder cancer, uninvestigated macroscopic haematuria
14. Women who are breastfeeding, pregnant or plan to get pregnant during the trial duration
15. Women of childbearing potential unwilling or unable to practice effective method of contraception
16. Participation in other clinical trials in the last month prior to baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2018-02-24 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
Absolute hearing improvement after 12 weeks | 12 weeks
  Absolute hearing improvement after 12 weeks measured with PTA using the mean value of the 3 most affected contiguous baseline frequencies (dB)

SECONDARY OUTCOMES:
complete hearing recovery after 12 weeks | 12 weeks
  Percentages of patients with complete hearing recovery after 12 weeks measured with PTA using the mean value of the 3 most affected contiguous frequencies at baseline

CONTACTS AND LOCATIONS:
Locations (3):
- Fakultni nemocnice Hradec Kralove, Hradec Králové, Czechia
- Universitätsklinik Freiburg, Freiburg im Breisgau, Germany
- Universitätsspital Zürich, Zurich, Switzerland